CLINICAL TRIAL: NCT06518486
Title: The Effectiveness of Foot-Ankle Exercise and Walking Exercise on Foot Neuropathy, Stress, Quality of Life, Blood Sugar Markers, Blood Pressure, Ankle-Brachial Index, and BMI Among Diabetes Mellitus Patients
Brief Title: Foot-Ankle Exercise and Walking Exercise on Diabetes Mellitus Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Siti Fadlilah, Principal Investigator, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RCT2024_Siti Fadlilah
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Foot; Diabetes Mellitus, Type 2; Diabetic Neuropathies; Diabetes Type 2; Diabetes; Diabetes Mellitus; Diabetes Complications
Keywords: Foot sensitivity; Stress; Quality of life; Fasting blood glucose; Body mass index; Blood pressure; Ankle-brachial index; Diabetes mellitus; Diabetic peripheral Neuropathies
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus, Type 2; Diabetic Neuropathies; Diabetes Mellitus; Diabetes Complications

STUDY DESIGN:
Intervention Model Description: Three arms parallel group design with 2 group interventions (foot-ankle exercise and walking exercise) and 1 control group
Who Masked: Outcomes Assessor
Masking Description: Data collectors who assess the outcomes and statistician who analyse the data are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Foot-ankle exercise group (Experimental): The group received intervention through health education, simulations, leaflets, and videos about foot-ankle exercise and practised independently for 12 weeks.
  Interventions: Other: Foot-ankle exercise
- Walking exercise group (Experimental): The group received intervention through health education, and leaflets about walking exercise and practised independently for 12 weeks.
  Interventions: Other: Walking exercise
- Control group (Active Comparator): The group that received intervention in the form of health education and leaflets about DM in general.
  Interventions: Other: Usual care and health education

INTERVENTIONS:
Other: Foot-ankle exercise — Foot-ankle exercise group will receive usual care provide by public health center and intervention through health education, leaflets, and videos about foot-ankle exercise. At the first meeting, participants will be taught how to do foot exercises and practice them in front of the instructor. Afterwards, participants will practice foot exercises independently without supervision for 12 weeks. One foot exercise session takes 10-15 minutes, while the physical activity target is for participants to fulfil a moderate level of physical activity (150 minutes/week). For this reason, participants are advised to do foot exercises for 2-3 sessions every day. The minimum duration of each session is 10 minutes, and two consecutive days without foot exercise are not allowed. Participants are asked to document all foot exercise practices in the logbook given at the first meeting. To monitor the intervention, we will contact participants by telephone for ±5 minutes/week.
  Arms: Foot-ankle exercise group
Other: Walking exercise — Participants in the walking exercise group will receive usual care provide by public health center and intervention through health education and leaflets about walking exercise. Participants will practice walking exercises independently without supervision for 12 weeks. Participants walked at the same speed as they did every day. The physical activity target to be achieved is for participants to be able to engage in a moderate level of physical activity (150 minutes/week). For this reason, participants are advised to do walking exercises with a minimum duration of 10 minutes for each session. Two consecutive days without walking exercise are not allowed, and a minimum of 150 minutes/week is allowed. Participants are asked to document all walking exercise practices in the logbook given at the first meeting. To monitor the intervention, we will contact participants by telephone for ±5 minutes/week.
  Arms: Walking exercise group
Other: Usual care and health education — Participants in the control group will receive the usual care provided by the community health center and intervention in the form of health education about DM in general.
  Arms: Control group

SUMMARY:
The primary purpose of this study is to determine the effectiveness of foot-ankle exercise and walking exercise on foot neuropathy, stress, and quality of life (QoL) among people with diabetes mellitus (PWDM). At the same time, the secondary purpose of this study is to determine the effectiveness of foot-ankle exercise and walking exercise on body mass index (BMI), fasting blood glucose (FBG), blood pressure (BP), and ankle-brachial index (ABI) among PWDM at baseline (before intervention/0 week), at 6-weeks and 12-weeks.

The research questions in this study include the following:

* Is foot-ankle exercise effective for foot neuropathy, stress, QoL, BMI, FBG, BP, and ABI for PWDM?
* Is walking exercise effective for foot neuropathy, stress, QoL, BMI, FBG, BP, and ABI for PWDM?
* Are there any differences in the mean scores of foot neuropathy, stress, QoL, BMI, FBG, BP, and ABI of PWDM within and between the foot-ankle exercise, walking exercise and control group at baseline, 6 weeks, and 12 weeks?
* Are there any mediators/moderators effect of BMI, FBG, blood pressure, ABI, and stress for influencing foot exercise and walking exercise interventions on foot neuropathy and QoL for PWDM?

Participants in the foot-ankle exercise group will be given health education about DM and foot-ankle exercise, as well as leaflets and videos. Participants will be taught how to practice foot-ankle exercises before the instructor. Afterwards, participants will practice foot-ankle exercises independently without supervision for 2-3 sessions every day for 12 weeks. Participants in the walking exercise group will be given health education about DM, walking exercises and leaflets. Participants will practice walking exercises independently without supervision for 12 weeks. Participants are advised to do walking exercises with a minimum duration of 10 minutes for each session and 150 minutes/week. Two consecutive days without walking exercise are not allowed. Participants in the control groups will be treated as active control and given health education on general DM topics and leaflets. All groups received usual care according to standards provided by public health services. Researchers will compare the groups to see the effect of the interventions on foot neuropathy, stress, QoL, BMI, FBG, BP, and ABI at three different time points: at baseline, 6 weeks, and 12 weeks.

DETAILED DESCRIPTION:
Intervention Development

This study focused on foot-ankle exercises modified from previous research and adapted to exercises developed by the Indonesian Endocrinology Association. Providing health education about DM in general and foot-ankle exercise is intended to increase participants' basic knowledge about DM and the importance of foot-ankle exercises. Foot-ankle exercise simulation and practice aim to ensure participants can do it well and independently. The leaflet contains the material presented during health education and is given to participants. A video was made containing the steps to do foot-ankle exercises. Researchers will upload videos of the foot-ankle exercises to YouTube. Participants will be given the video in soft file form and informed that they can access it via the researcher's YouTube channel. Walking exercises in this study adapted and modified from previous research. Providing health education about DM in general and walking exercises is intended to increase participants' basic knowledge about DM and the importance of walking exercise exercises. The leaflet contains the material presented during health education and is given to participants in walking exercise groups.

Content Validity

The content validity test in this study aims to validate the intervention procedures used during the research process. The details are: detail intervention of foot-ankle exercise and walking exercise, health education materials and leaflets for the control group, foot-ankle exercise groups, and walking exercise groups, videos of foot ankle exercises, standard operational procedures for measuring foot sensation and foot vibration, height and weight, BP, and ABI. The criteria for Experts: 1) Willing to be involved in the content validity study, 2) Doctor/nurse, 3) Have experience working in the clinical or research area on the topic of diabetes mellitus for more than 5 years. In this study, six experts are needed to achieve a content validation index (CVI) satisfaction of 0.83. Researchers will send formal invitations via email to experts. The files include an application letter, a cover letter containing the research objectives, expert panel criteria, intervention procedures to be assessed, and an assessment sheet. Assessment of each item uses a 1-4 Likert scale. Item with score <3 will be asked to provide comments or suggestions to help further refine the intervention protocol. Researchers will use item-level CVI (I-CVI) and the scale-level (S-CVI). The CVI value is satisfactory if I-CVI ≥0.80 and S-CVI ≥0.83. Items with a low CVI value will be revised according to the comments and suggestions of experts until the CVI value becomes satisfactory.

Participants Recruitment Process

Researchers will ask the District Health Service for information about public health centers (PHCs) with active Chronic Disease Management Program (PROLANIS) activities. Researchers will contact and collaborate with PHCs for participant recruitment. The research team will contact each potential participant and explain the research process. Researchers will also put-up posters in PHCs and also distribute these posters through social media. Potential participants willing to become participants can contact the contacts listed on the poster. For potential respondents who are willing, after signing the informed consent, they will be included in the chat group. Participants will be given a transportation fee of IDR 25,000 for each arrival during the data collection process.

Sample Size Calculation

Samples were calculated using G*Power sample size calculator v.3.1. using F test with an analysis of variance based on some criteria. Researchers will use small effect size (0.1), an α error probability of 0.05, and a power of 0.95; Number of groups 3 (foot-ankle exercise, walking exercise, and control group); and number of measurements 3 (baseline, 6-weeks, and 12 weeks). Based on the calculation, 312 participants were needed; and added an anticipated dropout of 20% (63 people), so the total sample size was 375. The total sample was divided into three groups; each group had 125 participants.

Randomization and Allocation Concealment

Eligible participants will be randomized by independent staff not involved in the recruitment and data collection process, with a ratio of 1:1:1 for each group. After baseline measurements, the randomization process will be carried out using the computer-generated randomization method. The method that will be used is random permuted blocks with size 3, 6, 9. The random numbers will be packaged in sequence, stored and locked in opaque envelopes to guarantee allocation concealment. This sequence will be kept private and stored in a place that assessors cannot access.

Intervention Delivery

Control group: The active control group was given health education on the topic of DM for 30 minutes and then given a leaflet.

Foot-ankle exercise group: Participants will be given health education on DM and foot-ankle exercise after the allocation procedure, followed by simulation and practice lasts 60 minutes. Participants were also given leaflets and videos to take home. Afterward, participants will practice independently without supervision for 12 weeks. Foot-ankle exercise consists of 10 movements. When doing foot exercises, participants sit comfortably without leaning, and the soles of their feet touch the floor and barefoot. These movements are:

A 1)Lift the soles of the feet with heels still touching the floor.2)Toes are bent to grip like chicken claws in this position.3)Repeat this movement 10x.

B 1)Lift the soles of the feet with heels still touching the floor. 2)Lower the soles of feet and raise heels with toes touching the floor. 3)Repeat this movement 10x.

C 1)Lift the soles of the feet with heels still touching the floor.2)Do circular movements from the inside to the outside for the soles of both feet.3)Repeat this movement 10x.

D 1)Lift the heels of both feet with toes still touching the floor.2)Do circular movements from the inside to the outside for the soles of both feet.3)Repeat this movement 10x.

E 1)Lift right knee and straighten it. The left leg remains in its original position.2)Move toes forward and backward.3)Repeat this movement 10x.4)Do the same for the left leg.

F 1)Lift right knee and straighten it.2)The left leg remains in its original position.3)Move toes towards face.4)Repeat this movement 10x.5)Do the same for the left leg.

G 1)Lift both knees of the right and left legs, then straighten them.2)Move toes towards face at the same time.3)Repeat this movement 10x.

H 1)Lift both knees of the right and left legs, then straighten them.2)Move both legs forward.3)Repeat this movement 10x.

I 1)Lift their right knee and straighten it. The left leg remains in its original position.2)Write the numbers 1-10 with feet.3)Do the same movement for the left leg.

J 1)Place newspapers as a base for the soles.2)Shape the newspaper into a ball using both feet.3)Open the newspaper ball again to become sheet-like before using both feet.4)Divide the newspaper into two parts using both feet.5)Tear one part of the newspaper into small pieces and collect it on top of the other part of the newspaper.6)The newspaper sheet containing small shreds is made into a ball using both feet.7)Throw the newspaper ball into the trash.

Walking exercise group: Participants will be given health education for 30 minutes, on DM and walking exercises and leaflet after the allocation procedure. Participants will practice walking exercises independently for 12 weeks.

Health education for all groups is provided by persons who have certificates as DM educators and carried out in subgroups with 7-10 members in each group. To avoid contamination, health education was implemented at different times, Fridays for control group, Saturday for foot-ankle exercise group, and Sunday for walking exercise group, with flexible implementation hours according to the agreement of each group. All group participants were included in the chat group (Whatsapp Messenger) so that researchers could communicate and monitor the implementation of the intervention.

Interventionist dan Outcome Investigators

Each research location has 1 health professional who carries out the intervention with criteria: having a master's degree in nursing, working as a health worker/health educator for at least 5 years, and having a certificate as a DM educator. Each research location has at least of 1 outcome investigator with the criteria of a health worker with a registration certificate.

Plan for Data Management/Analysis

Data analysis will use the intention to treat (ITT) principle. In addition, an analysis using the per-protocol (PP) principle will be carried out. Then, Researchers will compare the analysis results using ITT and PP and conduct a sensitivity test. The data analysis process uses the SPSS V.27 program. Researchers will conduct a normality test using the Kolmogorov Smirnov test; the data distribution is normal if the value is> 0.05. Researchers will use the Generalized Estimating Equation (GEE) test to analyze changes in outcomes between the foot-ankle exercise group vs control group, walking exercise group vs control group, and foot-ankle exercise group vs walking exercise group over time (baseline, six weeks, and 12 weeks). Baseline measurement and control group as reference. The significance value uses p value <0.05.

Comparison data of baseline respondents between the 3 groups for categorical data will be analyzed by the Chi-square/Fisher Exact test; for numerical data, ANOVA test for normal distributed or Friedman test for non-normally distributed. If a significant imbalance is found, an appropriate covariance adjustment analysis will be carried out in the data analysis. Analysis within group for each measurement time (baseline vs six weeks, baseline vs 12 weeks, six weeks vs 12 weeks) will use the Paired T-test if normally distributed or the Wilcoxon test if non-normally distributed. Meanwhile, the analysis between groups for each measurement time (T0, T1, and T2) will use the Independent T-test for normally distributed or the Mann-Whitney test for non-normally distributed.

Researchers will use path analysis to analyze the mediation/moderator of BMI, FBG, BP, ABI, and stress on the effects of foot-ankle exercise and walking exercise on foot sensitivity and QoL. The mediation analysis will use the bootstrap technique as a nonparametric procedure to test the statistical significance of various Partial Least Squares-Structural Equation Model (PLS-SEM) results, such as path coefficients. Researchers will use the software program SmartPLS 3 (SmartPLS GmbH, Bo¨nningstedt, Germany) to analyze the mediation effects. For PLS-SEM, Standard Root Mean Square Residual/SRMR can be used as a goodness-of-fit test to prevent model specification errors. SRMR is the difference between the observed correlation and the model's implied correlation matrix. As a result, it is possible to use the average magnitude of the difference between measured and predicted correlations as an absolute measure of (model) goodness-of-fit. A good fit is described as a value smaller than 0.10 or 0.08. The statistically significant level was set at 0.05 and 95% confidence intervals (CI) to test indirect effects. The result indicates a significant level if the 95% CI does not contain zero.

Monitor for Adverse Events

Adverse events that have the potential to occur include fatigue, muscle aches, pain and dizziness. Participants will record for themselves if adverse events occur and report to the team. The research team also monitored by telephone once a week, asking whether any adverse events had occurred and recording them. If excessive adverse events occur, investigators will immediately stop the intervention and carry out treatment.

ELIGIBILITY:
Inclusion Criteria:

* People with type 2 diabetes
* Aged 20-70 years
* Diagnosed with DM for at least 1 year
* Can walk without assistance
* Able to communicate well
* Can read and write
* Willing to be a respondent

Exclusion Criteria:

* Has a history of leg amputation
* Have a diagnosis of heart failure, kidney failure, pulmonary TB, stroke
* Patients with a history or under-treatment of mental disorders
* DM patients with foot ulcers
* DM patients with fractures or difficulty using the lower extremities

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2024-10-04 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Foot Neuropathy of People with Diabetes Mellitus | Baseline (before intervention/0 week), at 6-weeks and 12-weeks
  Foot neuropathy will be measured by MNSI. MNSI consist of MNSI-A (questionnaire) and MNSI-B (physical examination). Foot sensation will be measured using Semmes Weinstein Monofilament 10g. Participants will be given a stimulus for 1.5-2 seconds at 10 points on both legs. The locations are heel, dorsal surface of the foot (between the bases of 1st-2nd toes), toes (1st, 3rd, and 5th), metatarsal heads (1st, 3rd, 5th), and midfoot (medial and lateral). The results range from 0-10. Foot vibration measurement using Tunning Fork 128Hz. The vibrating TF will be placed on each leg in 4 locations (medial, malleolus, great toe, fifth toe). Participants were asked to feel the vibrations and signal by raising their hands if they were no longer felt. The observer will record the time from when the participant feels the initial until it disappears. The results consist of whether the participant felt the vibration or not (0-4) and the length of time participants can feel the vibration (in seconds).
Stress of People with Diabetes Mellitus | Baseline (before intervention/0 week), at 6-weeks and 12-weeks
  Stress will be measured using the Indonesian version of the Problem Areas in Diabetes (PAID) questionnaire. This study uses PAID Bahasa Indonesia, which we have previously tested for validity and reliability. PAID Bahasa Indonesia has 20 items and three factors, with a loading factor of 0.349-0.779 for each item. The results of exploratory factor analysis (EFA) and confirmatory factor analysis (CFA) show valid and reliable results. Cronbach's alpha for all items is 0.858, inter-class correlation 0.938, RMSEA=0.058, and SRMR=0.062. PAID Bahasa Indonesia consist of five answer choices using a Likert scale (0-4). The answer choice scores used were 'not a problem' (0), 'minor problem' (1), 'moderate problem' (2), 'somewhat serious problem' (3), and 'serious problem' (4). The total score ranged 0-80, with a higher score indicating greater stress.
Quality of Life of People with Diabetes Mellitus | Baseline (before intervention/0 week), at 6-weeks and 12-weeks
  QoL will be measured using the Indonesian version of the Diabetes Obstacles Questionnaire Short Version (DOQ-30) which we have previously tested for validity and reliability. DOQ-30 Bahasa Indonesia has nine factors and a 5-point Likert scale with answer options never (5), almost never (4), sometimes (3), often (2), and always (1). The total score ranges 30-150, with a higher score indicating a better QoL. Factors in the DOQ-30 are relationships with medical professionals, support from friends and family, knowledge of the disease, lifestyle changes, exercising, self-monitoring, uncertainty about a consultation, medication, and insulin use. EFA and CFA analysis showed valid and reliable results; Cronbach's alpha for all items was 0.930, and individual factors ranged from 0.730 to 0.848. The test-retest results were excellent (with interclass correlation coefficients of 0.910 to 0.973). The CFA test obtained RMSEA=0.057 and SRMR=0.067, indicating a good model fit.

SECONDARY OUTCOMES:
Fasting Blood Glucose (FBG) of People with Diabetes Mellitus | Baseline (before intervention/0 week), at 6-weeks and 12-weeks
  FBG were measured using venous blood after the respondent fasted for at least 8 hours. Blood analysis is carried out in the laboratory using the hexokinase enzymatic method. The researchers did not carry out this analysis, but they collaborated with the Independent Clinical Laboratory. All participants were measured according to standard operating procedures as a guide. The measurement results are documented in the observation sheet. The process of taking venous blood is carried out by nursing staff with the criteria of having a competency certificate and working for a minimum of 3 years.
Blood Pressure of People with Diabetes Mellitus | Baseline (before intervention/0 week), at 6-weeks and 12-weeks
  Blood pressure will be measured using a digital tensimeter, The Omron M3 Intellisense (Omron Healthcare Co Ltd), validated in previous research. Participants were asked to rest for at least 5 minutes before the measurement. Measurements were taken on the left arm in a sitting or supine position. Blood pressure consists of SBP and DBP in mmHg units. Then, the mean atrial pressure (MAP) will be calculated using the formula, MAP = DBP + 1/3(SBP - DBP) or MAP = DBP + 1/3(pulse pressure/PP) All participants were measured according to standard operating procedures as a guide. The measurement results are documented in the observation sheet.
Body Mass Index of People with Diabetes Mellitus | Baseline (before intervention/0 week), at 6-weeks and 12-weeks
  Participants were asked to stand up straight and remove footwear when their height and weight were checked. Body weight was measured using digital scales, and height using height-measuring devices. BMI is calculated using the formula body weight (kg) divided by height2 (m2). All participants were measured according to standard operating procedures as a guide. The measurement results are documented in the observation sheet.
Ankle-Brachial Index (ABI) of People with Diabetes Mellitus | Baseline (before intervention/0 week), at 6-weeks and 12-weeks
  ABI measurements will be carried out using continuous-wave Doppler ultrasound using SOPs prepared previously. Participants were asked to rest for at least 5 minutes, and measurements were taken in the supine position. BP was measured twice each at four locations: right arm, left arm, right leg and left leg. Arm blood pressure was measured by Doppler ultrasound in the humeral artery, while leg blood pressure was placed in the tibial artery. The cuff is inflated 20-30 mmHg and deflated slowly. The first sound heard is systolic blood pressure. The average blood pressure results from the two measurements at each location will be calculated to obtain the average blood pressure in the right arm, left arm, right leg and left leg. ABI will be calculated using the ankle SBP/brachial SBP formula. The results of these calculations produce the right and left ABI. The analysis will use the lowest ABI value between the two legs. The measurement results are documented in the observation sheet.
Adherence Participants in Experimental Group | 12-weeks
  The compliance of participants in both intervention groups in carrying out the program provided was measured using documentation from the logbook at the beginning of the meeting. The logbook contains information on the day, date, and time from start to finish, and it ends with the participant's signature.

CONTACTS AND LOCATIONS:
Overall Officials: Siti Fadlilah, Principal Investigator — Taipei Medical University
Locations (5):
- Indonesia (5):
  - Puskesmas Batang, Batang, Central Java
  - Puskesmas Musuk, Boyolali, Central Java
  - DPM Alexander, Sleman, Special Region of Yogyakarta
  - UPT Puskesmas Lunyuk, Sumbawa, West Nusa Tenggara
  - Puskesmas Kalasan, Sleman, Yogyakarta and West Nusa Tenggara

IPD SHARING:
Plan to Share IPD: Yes
Particular data will be shared: Individual participant data that underlie the results reported in this article after identification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 60 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose, for example, for a meta-analysis or other study.

REFERENCES:
- [Result] Herman WH, Pop-Busui R, Braffett BH, Martin CL, Cleary PA, Albers JW, Feldman EL; DCCT/EDIC Research Group. Use of the Michigan Neuropathy Screening Instrument as a measure of distal symmetrical peripheral neuropathy in Type 1 diabetes: results from the Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications. Diabet Med. 2012 Jul;29(7):937-44. doi: 10.1111/j.1464-5491.2012.03644.x. PMID 22417277
- [Result] Yang MC, Huang YY, Hsieh SH, Sun JH, Wang CC, Lin CH. Ankle-Brachial Index Is Independently Associated With Cardiovascular Outcomes and Foot Ulcers in Asian Patients With Type 2 Diabetes Mellitus. Front Endocrinol (Lausanne). 2021 Nov 18;12:752995. doi: 10.3389/fendo.2021.752995. eCollection 2021. PMID 34867797
- [Result] Welch GW, Jacobson AM, Polonsky WH. The Problem Areas in Diabetes Scale. An evaluation of its clinical utility. Diabetes Care. 1997 May;20(5):760-6. doi: 10.2337/diacare.20.5.760. PMID 9135939
- [Result] Weinstein AR, Sesso HD, Lee IM, Cook NR, Manson JE, Buring JE, Gaziano JM. Relationship of physical activity vs body mass index with type 2 diabetes in women. JAMA. 2004 Sep 8;292(10):1188-94. doi: 10.1001/jama.292.10.1188. PMID 15353531
- [Result] Tesfaye S, Boulton AJ, Dyck PJ, Freeman R, Horowitz M, Kempler P, Lauria G, Malik RA, Spallone V, Vinik A, Bernardi L, Valensi P; Toronto Diabetic Neuropathy Expert Group. Diabetic neuropathies: update on definitions, diagnostic criteria, estimation of severity, and treatments. Diabetes Care. 2010 Oct;33(10):2285-93. doi: 10.2337/dc10-1303. PMID 20876709
- [Result] Suryani M, Samekto W, Heri-Nugroho, Susanto H, Dwiantoro L. Effect of foot-ankle flexibility and resistance exercise in the secondary prevention of plantar foot diabetic ulcer. J Diabetes Complications. 2021 Sep;35(9):107968. doi: 10.1016/j.jdiacomp.2021.107968. Epub 2021 May 28. PMID 34187716
- [Result] Soleimani Tapehsari B, Alizadeh M, Khamseh ME, Seifouri S, Nojomi M. Physical Activity and Quality of Life in People with Type 2 Diabetes Mellitus: A Randomized Controlled Trial. Int J Prev Med. 2020 Jan 24;11:9. doi: 10.4103/ijpvm.IJPVM_202_18. eCollection 2020. PMID 32089809
- [Result] Diabetes Canada Clinical Practice Guidelines Expert Committee; Sigal RJ, Armstrong MJ, Bacon SL, Boule NG, Dasgupta K, Kenny GP, Riddell MC. Physical Activity and Diabetes. Can J Diabetes. 2018 Apr;42 Suppl 1:S54-S63. doi: 10.1016/j.jcjd.2017.10.008. No abstract available. PMID 29650112
- [Result] Shah SZA, Karam JA, Zeb A, Ullah R, Shah A, Haq IU, Ali I, Darain H, Chen H. Movement is Improvement: The Therapeutic Effects of Exercise and General Physical Activity on Glycemic Control in Patients with Type 2 Diabetes Mellitus: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Diabetes Ther. 2021 Mar;12(3):707-732. doi: 10.1007/s13300-021-01005-1. Epub 2021 Feb 5. PMID 33547579
- [Result] Schaper NC, van Netten JJ, Apelqvist J, Bus SA, Hinchliffe RJ, Lipsky BA; IWGDF Editorial Board. Practical Guidelines on the prevention and management of diabetic foot disease (IWGDF 2019 update). Diabetes Metab Res Rev. 2020 Mar;36 Suppl 1:e3266. doi: 10.1002/dmrr.3266. PMID 32176447
- [Result] Park S, Kim J, Lee J. Effects of Exercise Intervention on Adults With Both Hypertension and Type 2 Diabetes Mellitus: A Systematic Review and Meta-analysis. J Cardiovasc Nurs. 2021 Jan/Feb;36(1):23-33. doi: 10.1097/JCN.0000000000000651. PMID 32011348
- [Result] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c869. doi: 10.1136/bmj.c869. No abstract available. PMID 20332511
- [Result] Rac-Albu M, Iliuta L, Guberna SM, Sinescu C. The role of ankle-brachial index for predicting peripheral arterial disease. Maedica (Bucur). 2014 Sep;9(3):295-302. PMID 25705296
- [Result] Lu B, Hu J, Wen J, Zhang Z, Zhou L, Li Y, Hu R. Determination of peripheral neuropathy prevalence and associated factors in Chinese subjects with diabetes and pre-diabetes - ShangHai Diabetic neuRopathy Epidemiology and Molecular Genetics Study (SH-DREAMS). PLoS One. 2013 Apr 16;8(4):e61053. doi: 10.1371/journal.pone.0061053. Print 2013. PMID 23613782
- [Result] Kirwan JP, Sacks J, Nieuwoudt S. The essential role of exercise in the management of type 2 diabetes. Cleve Clin J Med. 2017 Jul;84(7 Suppl 1):S15-S21. doi: 10.3949/ccjm.84.s1.03. PMID 28708479
- [Result] Kelley GA, Kelley KS. Progressive resistance exercise and resting blood pressure : A meta-analysis of randomized controlled trials. Hypertension. 2000 Mar;35(3):838-43. doi: 10.1161/01.hyp.35.3.838. PMID 10720604
- [Result] Karstoft K, Clark MA, Jakobsen I, Muller IA, Pedersen BK, Solomon TP, Ried-Larsen M. The effects of 2 weeks of interval vs continuous walking training on glycaemic control and whole-body oxidative stress in individuals with type 2 diabetes: a controlled, randomised, crossover trial. Diabetologia. 2017 Mar;60(3):508-517. doi: 10.1007/s00125-016-4170-6. Epub 2016 Dec 9. PMID 27942800
- [Result] Kanchanasamut W, Pensri P. Effects of weight-bearing exercise on a mini-trampoline on foot mobility, plantar pressure and sensation of diabetic neuropathic feet; a preliminary study. Diabet Foot Ankle. 2017 Feb 20;8(1):1287239. doi: 10.1080/2000625X.2017.1287239. eCollection 2017. PMID 28326159
- [Result] Kanade RV, van Deursen RW, Harding K, Price P. Walking performance in people with diabetic neuropathy: benefits and threats. Diabetologia. 2006 Aug;49(8):1747-54. doi: 10.1007/s00125-006-0309-1. Epub 2006 Jun 7. PMID 16758177
- [Result] Hoogendoorn SW, Rutten GEHM, Hart HE, de Wolf C, Vos RC. A simple to implement and low-cost supervised walking programme in highly motivated individuals with or at risk for type 2 diabetes: An observational study with a pre-post design. Prev Med Rep. 2018 Nov 7;13:30-36. doi: 10.1016/j.pmedr.2018.11.003. eCollection 2019 Mar. PMID 30510891
- [Result] Henderson AD, Johnson AW, Rasmussen LG, Peine WP, Symons SH, Scoresby KA, Ridge ST, Bruening DA. Early-Stage Diabetic Neuropathy Reduces Foot Strength and Intrinsic but Not Extrinsic Foot Muscle Size. J Diabetes Res. 2020 Mar 12;2020:9536362. doi: 10.1155/2020/9536362. eCollection 2020. PMID 32258170
- [Result] Gray N, Picone G, Sloan F, Yashkin A. Relation between BMI and diabetes mellitus and its complications among US older adults. South Med J. 2015 Jan;108(1):29-36. doi: 10.14423/SMJ.0000000000000214. PMID 25580754
- [Result] Gram B, Christensen R, Christiansen C, Gram J. Effects of nordic walking and exercise in type 2 diabetes mellitus: a randomized controlled trial. Clin J Sport Med. 2010 Sep;20(5):355-61. doi: 10.1227/NEU.0b013e3181e56e0a. PMID 20818193
- [Result] Ferrannini E, Cushman WC. Diabetes and hypertension: the bad companions. Lancet. 2012 Aug 11;380(9841):601-10. doi: 10.1016/S0140-6736(12)60987-8. PMID 22883509
- [Result] Dong XL, Guan F, Xu SJ, Zhu LX, Zhang PP, Cheng AB, Liu TJ. Influence of blood glucose level on the prognosis of patients with diabetes mellitus complicated with ischemic stroke. J Res Med Sci. 2018 Jan 29;23:10. doi: 10.4103/1735-1995.223951. eCollection 2018. PMID 29456567
- [Result] Defay R, Delcourt C, Ranvier M, Lacroux A, Papoz L. Relationships between physical activity, obesity and diabetes mellitus in a French elderly population: the POLA study. Pathologies Oculaires liees a l' Age. Int J Obes Relat Metab Disord. 2001 Apr;25(4):512-8. doi: 10.1038/sj.ijo.0801570. PMID 11319655
- [Result] de Boer IH, Bangalore S, Benetos A, Davis AM, Michos ED, Muntner P, Rossing P, Zoungas S, Bakris G. Diabetes and Hypertension: A Position Statement by the American Diabetes Association. Diabetes Care. 2017 Sep;40(9):1273-1284. doi: 10.2337/dci17-0026. No abstract available. PMID 28830958
- [Result] Cruvinel-Junior RH, Ferreira JSSP, Verissimo JL, Monteiro RL, Suda EY, Silva EQ, Sacco ICN. Could an Internet-Based Foot-Ankle Therapeutic Exercise Program Modify Clinical Outcomes and Gait Biomechanics in People with Diabetic Neuropathy? A Clinical Proof-of-Concept Study. Sensors (Basel). 2022 Dec 7;22(24):9582. doi: 10.3390/s22249582. PMID 36559949
- [Result] Crawford F, Inkster M, Kleijnen J, Fahey T. Predicting foot ulcers in patients with diabetes: a systematic review and meta-analysis. QJM. 2007 Feb;100(2):65-86. doi: 10.1093/qjmed/hcl140. PMID 17277315
- [Result] Cho NH, Shaw JE, Karuranga S, Huang Y, da Rocha Fernandes JD, Ohlrogge AW, Malanda B. IDF Diabetes Atlas: Global estimates of diabetes prevalence for 2017 and projections for 2045. Diabetes Res Clin Pract. 2018 Apr;138:271-281. doi: 10.1016/j.diabres.2018.02.023. Epub 2018 Feb 26. PMID 29496507
- [Result] Childs E, de Wit H. Regular exercise is associated with emotional resilience to acute stress in healthy adults. Front Physiol. 2014 May 1;5:161. doi: 10.3389/fphys.2014.00161. eCollection 2014. PMID 24822048
- [Result] Cai H, Li G, Zhang P, Xu D, Chen L. Effect of exercise on the quality of life in type 2 diabetes mellitus: a systematic review. Qual Life Res. 2017 Mar;26(3):515-530. doi: 10.1007/s11136-016-1481-5. Epub 2016 Dec 18. PMID 27990609
- [Result] Bus SA, Lavery LA, Monteiro-Soares M, Rasmussen A, Raspovic A, Sacco ICN, van Netten JJ; International Working Group on the Diabetic Foot. Guidelines on the prevention of foot ulcers in persons with diabetes (IWGDF 2019 update). Diabetes Metab Res Rev. 2020 Mar;36 Suppl 1:e3269. doi: 10.1002/dmrr.3269. PMID 32176451
- [Result] Boulton AJ, Vileikyte L, Ragnarson-Tennvall G, Apelqvist J. The global burden of diabetic foot disease. Lancet. 2005 Nov 12;366(9498):1719-24. doi: 10.1016/S0140-6736(05)67698-2. PMID 16291066
- [Result] Bonora E, Trombetta M, Dauriz M, Travia D, Cacciatori V, Brangani C, Negri C, Perrone F, Pichiri I, Stoico V, Zoppini G, Rinaldi E, Da Prato G, Boselli ML, Santi L, Moschetta F, Zardini M, Bonadonna RC. Chronic complications in patients with newly diagnosed type 2 diabetes: prevalence and related metabolic and clinical features: the Verona Newly Diagnosed Type 2 Diabetes Study (VNDS) 9. BMJ Open Diabetes Res Care. 2020 Aug;8(1):e001549. doi: 10.1136/bmjdrc-2020-001549. PMID 32819978
- [Result] Birke JA, Patout CA Jr, Foto JG. Factors associated with ulceration and amputation in the neuropathic foot. J Orthop Sports Phys Ther. 2000 Feb;30(2):91-7. doi: 10.2519/jospt.2000.30.2.91. PMID 10693087
- [Result] Asmar R, Khabouth J, Topouchian J, El Feghali R, Mattar J. Validation of three automatic devices for self-measurement of blood pressure according to the International Protocol: The Omron M3 Intellisense (HEM-7051-E), the Omron M2 Compact (HEM 7102-E), and the Omron R3-I Plus (HEM 6022-E). Blood Press Monit. 2010 Feb;15(1):49-54. doi: 10.1097/MBP.0b013e3283354b11. PMID 20032779
- [Result] Asfaw MS, Dagne WK. Physical activity can improve diabetes patients' glucose control; A systematic review and meta-analysis. Heliyon. 2022 Dec 13;8(12):e12267. doi: 10.1016/j.heliyon.2022.e12267. eCollection 2022 Dec. PMID 36578408
- [Result] Alves-Cabratosa L, Comas-Cufi M, Ponjoan A, Garcia-Gil M, Marti-Lluch R, Blanch J, Elosua-Bayes M, Parramon D, Camos L, Guzman L, Ramos R. Levels of ankle-brachial index and the risk of diabetes mellitus complications. BMJ Open Diabetes Res Care. 2020 Mar;8(1):e000977. doi: 10.1136/bmjdrc-2019-000977. PMID 32144131
- [Result] Alqahtani KM, Bhangoo M, Vaida F, Denenberg JO, Allison MA, Criqui MH. Predictors of Change in the Ankle Brachial Index with Exercise. Eur J Vasc Endovasc Surg. 2018 Mar;55(3):399-404. doi: 10.1016/j.ejvs.2017.12.004. Epub 2018 Jan 20. PMID 29371037
- [Result] Barone Gibbs B, Dobrosielski DA, Althouse AD, Stewart KJ. The effect of exercise training on ankle-brachial index in type 2 diabetes. Atherosclerosis. 2013 Sep;230(1):125-30. doi: 10.1016/j.atherosclerosis.2013.07.002. Epub 2013 Jul 14. PMID 23958264
- [Result] Aboyans V, Criqui MH, Abraham P, Allison MA, Creager MA, Diehm C, Fowkes FG, Hiatt WR, Jonsson B, Lacroix P, Marin B, McDermott MM, Norgren L, Pande RL, Preux PM, Stoffers HE, Treat-Jacobson D; American Heart Association Council on Peripheral Vascular Disease; Council on Epidemiology and Prevention; Council on Clinical Cardiology; Council on Cardiovascular Nursing; Council on Cardiovascular Radiology and Intervention, and Council on Cardiovascular Surgery and Anesthesia. Measurement and interpretation of the ankle-brachial index: a scientific statement from the American Heart Association. Circulation. 2012 Dec 11;126(24):2890-909. doi: 10.1161/CIR.0b013e318276fbcb. Epub 2012 Nov 16. No abstract available. PMID 23159553
- [Result] Adu MD, Malabu UH, Malau-Aduli AEO, Malau-Aduli BS. Enablers and barriers to effective diabetes self-management: A multi-national investigation. PLoS One. 2019 Jun 5;14(6):e0217771. doi: 10.1371/journal.pone.0217771. eCollection 2019. PMID 31166971
- [Result] Aloke C, Egwu CO, Aja PM, Obasi NA, Chukwu J, Akumadu BO, Ogbu PN, Achilonu I. Current Advances in the Management of Diabetes Mellitus. Biomedicines. 2022 Sep 29;10(10):2436. doi: 10.3390/biomedicines10102436. PMID 36289697
- [Result] American Diabetes Association. Standards of medical care in diabetes-2015 abridged for primary care providers. Clin Diabetes. 2015 Apr;33(2):97-111. doi: 10.2337/diaclin.33.2.97. No abstract available. PMID 25897193
- [Result] American Diabetes Association. 2. Classification and Diagnosis of Diabetes: Standards of Medical Care in Diabetes-2021. Diabetes Care. 2021 Jan;44(Suppl 1):S15-S33. doi: 10.2337/dc21-S002. PMID 33298413
- [Result] Amin N, Doupis J. Diabetic foot disease: From the evaluation of the "foot at risk" to the novel diabetic ulcer treatment modalities. World J Diabetes. 2016 Apr 10;7(7):153-64. doi: 10.4239/wjd.v7.i7.153. PMID 27076876
- [Result] Aschalew AY, Yitayal M, Minyihun A. Health-related quality of life and associated factors among patients with diabetes mellitus at the University of Gondar referral hospital. Health Qual Life Outcomes. 2020 Mar 10;18(1):62. doi: 10.1186/s12955-020-01311-5. PMID 32156282
- [Result] Aylin K, Arzu D, Sabri S, Handan TE, Ridvan A. The effect of combined resistance and home-based walking exercise in type 2 diabetes patients. Int J Diabetes Dev Ctries. 2009 Oct;29(4):159-65. doi: 10.4103/0973-3930.57347. PMID 20336198
- [Result] Battista F, Ermolao A, van Baak MA, Beaulieu K, Blundell JE, Busetto L, Carraca EV, Encantado J, Dicker D, Farpour-Lambert N, Pramono A, Bellicha A, Oppert JM. Effect of exercise on cardiometabolic health of adults with overweight or obesity: Focus on blood pressure, insulin resistance, and intrahepatic fat-A systematic review and meta-analysis. Obes Rev. 2021 Jul;22 Suppl 4(Suppl 4):e13269. doi: 10.1111/obr.13269. Epub 2021 May 6. PMID 33960110
- [Result] Belli T, Ribeiro LF, Ackermann MA, Baldissera V, Gobatto CA, Galdino da Silva R. Effects of 12-week overground walking training at ventilatory threshold velocity in type 2 diabetic women. Diabetes Res Clin Pract. 2011 Sep;93(3):337-43. doi: 10.1016/j.diabres.2011.05.007. Epub 2011 Jun 1. PMID 21636159
- [Result] Boulton AJ, Vinik AI, Arezzo JC, Bril V, Feldman EL, Freeman R, Malik RA, Maser RE, Sosenko JM, Ziegler D; American Diabetes Association. Diabetic neuropathies: a statement by the American Diabetes Association. Diabetes Care. 2005 Apr;28(4):956-62. doi: 10.2337/diacare.28.4.956. No abstract available. PMID 15793206
- [Result] Brown SJ, Handsaker JC, Bowling FL, Boulton AJ, Reeves ND. Diabetic peripheral neuropathy compromises balance during daily activities. Diabetes Care. 2015 Jun;38(6):1116-22. doi: 10.2337/dc14-1982. Epub 2015 Mar 12. PMID 25765355
- [Result] Bull FC, Al-Ansari SS, Biddle S, Borodulin K, Buman MP, Cardon G, Carty C, Chaput JP, Chastin S, Chou R, Dempsey PC, DiPietro L, Ekelund U, Firth J, Friedenreich CM, Garcia L, Gichu M, Jago R, Katzmarzyk PT, Lambert E, Leitzmann M, Milton K, Ortega FB, Ranasinghe C, Stamatakis E, Tiedemann A, Troiano RP, van der Ploeg HP, Wari V, Willumsen JF. World Health Organization 2020 guidelines on physical activity and sedentary behaviour. Br J Sports Med. 2020 Dec;54(24):1451-1462. doi: 10.1136/bjsports-2020-102955. PMID 33239350
- [Result] Cerrahoglu L, Kosan U, Sirin TC, Ulusoy A. Range of Motion and Plantar Pressure Evaluation for the Effects of Self-Care Foot Exercises on Diabetic Patients with and Without Neuropathy. J Am Podiatr Med Assoc. 2016 May;106(3):189-200. doi: 10.7547/14-095. PMID 27269974
- [Result] Colberg SR, Sigal RJ, Yardley JE, Riddell MC, Dunstan DW, Dempsey PC, Horton ES, Castorino K, Tate DF. Physical Activity/Exercise and Diabetes: A Position Statement of the American Diabetes Association. Diabetes Care. 2016 Nov;39(11):2065-2079. doi: 10.2337/dc16-1728. No abstract available. PMID 27926890
- [Result] Ankle Brachial Index Collaboration; Fowkes FG, Murray GD, Butcher I, Heald CL, Lee RJ, Chambless LE, Folsom AR, Hirsch AT, Dramaix M, deBacker G, Wautrecht JC, Kornitzer M, Newman AB, Cushman M, Sutton-Tyrrell K, Fowkes FG, Lee AJ, Price JF, d'Agostino RB, Murabito JM, Norman PE, Jamrozik K, Curb JD, Masaki KH, Rodriguez BL, Dekker JM, Bouter LM, Heine RJ, Nijpels G, Stehouwer CD, Ferrucci L, McDermott MM, Stoffers HE, Hooi JD, Knottnerus JA, Ogren M, Hedblad B, Witteman JC, Breteler MM, Hunink MG, Hofman A, Criqui MH, Langer RD, Fronek A, Hiatt WR, Hamman R, Resnick HE, Guralnik J, McDermott MM. Ankle brachial index combined with Framingham Risk Score to predict cardiovascular events and mortality: a meta-analysis. JAMA. 2008 Jul 9;300(2):197-208. doi: 10.1001/jama.300.2.197. PMID 18612117
- [Result] Craig AB, Strauss MB, Daniller A, Miller SS. Foot sensation testing in the patient with diabetes: introduction of the quick & easy assessment tool. Wounds. 2014 Aug;26(8):221-31. PMID 25860638
- [Result] de la Vega R, Jimenez-Castuera R, Leyton-Roman M. Impact of Weekly Physical Activity on Stress Response: An Experimental Study. Front Psychol. 2021 Jan 12;11:608217. doi: 10.3389/fpsyg.2020.608217. eCollection 2020. PMID 33510685
- [Result] Dube S, Hulke SM, Wakode SL, Khadanga S, Thakare AE, Bharshankar RN, Pakhare A. Effectiveness of Semmes Weinstein 10 gm monofilament in diabetic peripheral neuropathy taking nerve conduction and autonomic function study as reference tests. J Family Med Prim Care. 2022 Oct;11(10):6204-6208. doi: 10.4103/jfmpc.jfmpc_195_22. Epub 2022 Oct 31. PMID 36618173
- [Result] Faizah R, Efendi F, Suprajitno S. The effects of foot exercise with audiovisual and group support foot exercises to diabetes mellitus patients. J Diabetes Metab Disord. 2021 Feb 22;20(1):377-382. doi: 10.1007/s40200-021-00756-9. eCollection 2021 Jun. PMID 34178845
- [Result] Ferreira JSSP, Sacco ICN, Siqueira AA, Almeida MHM, Sartor CD. Rehabilitation technology for self-care: Customised foot and ankle exercise software for people with diabetes. PLoS One. 2019 Jun 20;14(6):e0218560. doi: 10.1371/journal.pone.0218560. eCollection 2019. PMID 31220155
- [Result] Francia P, Anichini R, De Bellis A, Seghieri G, Lazzeri R, Paternostro F, Gulisano M. Diabetic foot prevention: the role of exercise therapy in the treatment of limited joint mobility, muscle weakness and reduced gait speed. Ital J Anat Embryol. 2015;120(1):21-32. PMID 26738255
- [Result] Guglani R, Shenoy S, Sandhu JS. Effect of progressive pedometer based walking intervention on quality of life and general well being among patients with type 2 diabetes. J Diabetes Metab Disord. 2014 Nov 29;13(1):110. doi: 10.1186/s40200-014-0110-5. eCollection 2014. PMID 25493265
- [Result] Hyun S, Forbang NI, Allison MA, Denenberg JO, Criqui MH, Ix JH. Ankle-brachial index, toe-brachial index, and cardiovascular mortality in persons with and without diabetes mellitus. J Vasc Surg. 2014 Aug;60(2):390-5. doi: 10.1016/j.jvs.2014.02.008. Epub 2014 Mar 21. PMID 24657294
- [Result] Ingrosso DMF, Primavera M, Samvelyan S, Tagi VM, Chiarelli F. Stress and Diabetes Mellitus: Pathogenetic Mechanisms and Clinical Outcome. Horm Res Paediatr. 2023;96(1):34-43. doi: 10.1159/000522431. Epub 2022 Feb 4. PMID 35124671
- [Result] Inzucchi SE, Bergenstal RM, Buse JB, Diamant M, Ferrannini E, Nauck M, Peters AL, Tsapas A, Wender R, Matthews DR. Management of hyperglycemia in type 2 diabetes, 2015: a patient-centered approach: update to a position statement of the American Diabetes Association and the European Association for the Study of Diabetes. Diabetes Care. 2015 Jan;38(1):140-9. doi: 10.2337/dc14-2441. No abstract available. PMID 25538310
- [Result] Islam FMA, Islam MA, Hosen MA, Lambert EA, Maddison R, Lambert GW, Thompson BR. Associations of physical activity levels, and attitudes towards physical activity with blood pressure among adults with high blood pressure in Bangladesh. PLoS One. 2023 Feb 3;18(2):e0280879. doi: 10.1371/journal.pone.0280879. eCollection 2023. PMID 36735692
- [Result] Kirwan JP, Solomon TP, Wojta DM, Staten MA, Holloszy JO. Effects of 7 days of exercise training on insulin sensitivity and responsiveness in type 2 diabetes mellitus. Am J Physiol Endocrinol Metab. 2009 Jul;297(1):E151-6. doi: 10.1152/ajpendo.00210.2009. Epub 2009 Apr 21. PMID 19383872
- [Result] Lee S, Kim H, Choi S, Park Y, Kim Y, Cho B. Clinical usefulness of the two-site Semmes-Weinstein monofilament test for detecting diabetic peripheral neuropathy. J Korean Med Sci. 2003 Feb;18(1):103-7. doi: 10.3346/jkms.2003.18.1.103. PMID 12589096
- [Result] Lin X, Xu Y, Pan X, Xu J, Ding Y, Sun X, Song X, Ren Y, Shan PF. Global, regional, and national burden and trend of diabetes in 195 countries and territories: an analysis from 1990 to 2025. Sci Rep. 2020 Sep 8;10(1):14790. doi: 10.1038/s41598-020-71908-9. PMID 32901098
- [Result] Linderman GC, Lu J, Lu Y, Sun X, Xu W, Nasir K, Schulz W, Jiang L, Krumholz HM. Association of Body Mass Index With Blood Pressure Among 1.7 Million Chinese Adults. JAMA Netw Open. 2018 Aug 3;1(4):e181271. doi: 10.1001/jamanetworkopen.2018.1271. PMID 30646115
- [Result] Monteiro RL, Ferreira JSSP, Silva EQ, Cruvinel-Junior RH, Verissimo JL, Bus SA, Sacco ICN. Foot-ankle therapeutic exercise program can improve gait speed in people with diabetic neuropathy: a randomized controlled trial. Sci Rep. 2022 May 9;12(1):7561. doi: 10.1038/s41598-022-11745-0. PMID 35534614
- [Result] Oluchi SE, Manaf RA, Ismail S, Kadir Shahar H, Mahmud A, Udeani TK. Health Related Quality of Life Measurements for Diabetes: A Systematic Review. Int J Environ Res Public Health. 2021 Sep 1;18(17):9245. doi: 10.3390/ijerph18179245. PMID 34501838
- [Result] Pilv L, Vermeire E, Ratsep A, Moreau A, Nikolic D, Petek D, Yaman H, Oona M, Kalda R. Development and validation of the short version of the diabetes obstacles questionnaire (DOQ-30) in six European countries. Eur J Gen Pract. 2016;22(1):16-22. doi: 10.3109/13814788.2015.1093619. Epub 2015 Nov 18. PMID 26578192
- [Result] Polonsky WH, Anderson BJ, Lohrer PA, Welch G, Jacobson AM, Aponte JE, Schwartz CE. Assessment of diabetes-related distress. Diabetes Care. 1995 Jun;18(6):754-60. doi: 10.2337/diacare.18.6.754. PMID 7555499
- [Result] Qiu S, Cai X, Schumann U, Velders M, Sun Z, Steinacker JM. Impact of walking on glycemic control and other cardiovascular risk factors in type 2 diabetes: a meta-analysis. PLoS One. 2014 Oct 17;9(10):e109767. doi: 10.1371/journal.pone.0109767. eCollection 2014. PMID 25329391
- [Result] Rias YA, Kurniawan AL, Chang CW, Gordon CJ, Tsai HT. Synergistic Effects of Regular Walking and Alkaline Electrolyzed Water on Decreasing Inflammation and Oxidative Stress, and Increasing Quality of Life in Individuals with Type 2 Diabetes: A Community Based Randomized Controlled Trial. Antioxidants (Basel). 2020 Oct 1;9(10):946. doi: 10.3390/antiox9100946. PMID 33019646
- [Result] Saeedi P, Petersohn I, Salpea P, Malanda B, Karuranga S, Unwin N, Colagiuri S, Guariguata L, Motala AA, Ogurtsova K, Shaw JE, Bright D, Williams R; IDF Diabetes Atlas Committee. Global and regional diabetes prevalence estimates for 2019 and projections for 2030 and 2045: Results from the International Diabetes Federation Diabetes Atlas, 9th edition. Diabetes Res Clin Pract. 2019 Nov;157:107843. doi: 10.1016/j.diabres.2019.107843. Epub 2019 Sep 10. PMID 31518657
- [Result] Sartor CD, Hasue RH, Cacciari LP, Butugan MK, Watari R, Passaro AC, Giacomozzi C, Sacco IC. Effects of strengthening, stretching and functional training on foot function in patients with diabetic neuropathy: results of a randomized controlled trial. BMC Musculoskelet Disord. 2014 Apr 27;15:137. doi: 10.1186/1471-2474-15-137. PMID 24767584
- [Result] Takahara M, Fujiwara Y, Sakamoto F, Katakami N, Matsuoka TA, Kaneto H, Shimomura I. Assessment of vibratory sensation with a tuning fork at different sites in Japanese patients with diabetes mellitus. J Diabetes Investig. 2014 Feb 12;5(1):90-3. doi: 10.1111/jdi.12126. Epub 2013 Aug 28. PMID 24843743
- [Result] Tan LS. The clinical use of the 10g monofilament and its limitations: a review. Diabetes Res Clin Pract. 2010 Oct;90(1):1-7. doi: 10.1016/j.diabres.2010.06.021. Epub 2010 Jul 22. PMID 20655123
- [Result] Umpierre D, Ribeiro PA, Kramer CK, Leitao CB, Zucatti AT, Azevedo MJ, Gross JL, Ribeiro JP, Schaan BD. Physical activity advice only or structured exercise training and association with HbA1c levels in type 2 diabetes: a systematic review and meta-analysis. JAMA. 2011 May 4;305(17):1790-9. doi: 10.1001/jama.2011.576. PMID 21540423
- [Result] Wang Y, Mou Q, Zhao D, Xu Y, Hu D, Ma H, Liu J, Guo X, Li J. Predictive value of ankle-brachial index and blood glucose on the outcomes of six-year all-cause mortality and cardiovascular mortality in a Chinese population of type 2 diabetes patients. Int Angiol. 2012 Dec;31(6):586-94. PMID 23222938
- [Result] Whelton SP, Chin A, Xin X, He J. Effect of aerobic exercise on blood pressure: a meta-analysis of randomized, controlled trials. Ann Intern Med. 2002 Apr 2;136(7):493-503. doi: 10.7326/0003-4819-136-7-200204020-00006. PMID 11926784
- [Result] Win MMTM, Fukai K, Nyunt HH, Linn KZ. Hand and foot exercises for diabetic peripheral neuropathy: A randomized controlled trial. Nurs Health Sci. 2020 Jun;22(2):416-426. doi: 10.1111/nhs.12676. Epub 2019 Dec 26. PMID 31876991
- [Result] Young MJ, Breddy JL, Veves A, Boulton AJ. The prediction of diabetic neuropathic foot ulceration using vibration perception thresholds. A prospective study. Diabetes Care. 1994 Jun;17(6):557-60. doi: 10.2337/diacare.17.6.557. PMID 8082524
- [Result] Yuenyongchaiwat K, Pipatsitipong D, Sangprasert P. Increasing walking steps daily can reduce blood pressure and diabetes in overweight participants. Diabetol Int. 2017 Aug 7;9(1):75-79. doi: 10.1007/s13340-017-0333-z. eCollection 2018 Feb. PMID 30603352
- [Result] Zheng ZJ, Rosamond WD, Chambless LE, Nieto FJ, Barnes RW, Hutchinson RG, Tyroler HA, Heiss G; ARIC Investigators. Lower extremity arterial disease assessed by ankle-brachial index in a middle-aged population of African Americans and whites: the Atherosclerosis Risk in Communities (ARIC) Study. Am J Prev Med. 2005 Dec;29(5 Suppl 1):42-9. doi: 10.1016/j.amepre.2005.07.019. PMID 16389125
- [Result] Zhu X, Zhao L, Chen J, Lin C, Lv F, Hu S, Cai X, Zhang L, Ji L. The Effect of Physical Activity on Glycemic Variability in Patients With Diabetes: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Front Endocrinol (Lausanne). 2021 Nov 17;12:767152. doi: 10.3389/fendo.2021.767152. eCollection 2021. PMID 34867812
- See also: International Diabetes Federation, I. (2021). IDF Diabetes Atlas 10th edition. — http://www.diabetesatlas.org